CLINICAL TRIAL: NCT03380286
Title: Evaluation of Effectiveness and Safety of Firehawk® Stent in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: IRIS-Firehawk® Cohort in the IRIS-DES Registry
Acronym: IRIS Firehawk
Status: Withdrawn | Type: Observational
Why Stopped: Funding issue
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Professor, Division of Cardiology, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2017-09
Record Dates: First submitted 2017-12-17; First posted 2017-12-21 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Coronary Stenosis; Coronary Disease
Keywords: Firehawk; Coronary Artery Disease; Drug Eluting Stent
MeSH Terms: conditions — Coronary Stenosis; Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Stenosis
  Interventions: Device: Firehawk

INTERVENTIONS:
Device: Firehawk — Firehawk stent

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of Firehawk® stent in the "real world" daily practice as compared with other drug-eluting stents.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Patient with Firehawk® coronary stent

Exclusion Criteria:

* Intervention with Firehawk® coronary stent and other drug eluting stent at the same time
* Life-expectancy less than 1 year
* Cardiac shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Firehawk® coronary stent
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite event rate of death, non-fatal myocardial infarction (MI), or Target- Vessel Revascularization (TVR) | 1 year

SECONDARY OUTCOMES:
All cause death | 5 year
Cardiac death | 5 year
Myocardial Infarction | 5 year
Composite event rate of death or myocardial infarction (MI) | 5 year
Composite event rate of cardiac death or myocardial infarction (MI) | 5 year
Target- Vessel Revascularization | 5 year
Target- Lesion Revascularization | 5 year
Stent thrombosis | 5 year
Procedural Success rate | 5 year
  Procedural success rate is defined as < 30% final stenosis and the absence of in-hospital event including death, Q wave myocardial infarction, urgent repeat revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided